CLINICAL TRIAL: NCT01045655
Title: For Moms: Culturally Relevant Treatment Services for Perinatal Depression
Brief Title: MOMCare: Culturally Relevant Treatment Services for Perinatal Depression
Acronym: MOMCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nancy Grote, Research Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH084897 (NIH); R01MH084897 (NIH)
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Depression
Keywords: Depression; Perinatal care; Postpartum period; Pregnancy; Female; Low-income population
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MOMCare intervention (Experimental): Depression care treatment with study depression care specialist (brief interpersonal psychotherapy or pharmacotherapy)
  Interventions: Behavioral: MOMCare
- Care Plus (No Intervention): Usual care group; referral to community mental health treatment

INTERVENTIONS:
Behavioral: MOMCare — 8 sessions of brief interpersonal psychotherapy or medication management; maintenance sessions through 12 months postpartum.
  Arms: MOMCare intervention

SUMMARY:
The study will evaluate the effectiveness of a culturally relevant, multi-component intervention for antenatal depression. The intervention includes an engagement session, and the woman's choice of brief interpersonal psychotherapy and/or pharmacotherapy in a stepped care treatment for depression model.

DETAILED DESCRIPTION:
The randomized control trial will evaluate the effects of a culturally relevant, multi-component intervention for antenatal depression. MOMCare has the potential to overcome patient, provider, and system-level barriers to care and engage depressed, low-income women in evidence-based treatments to reduce antenatal depressive symptoms, improve maternal psychosocial functioning, and ameliorate postpartum depression. Specific Aim 1: To evaluate the impact of MOMCare on treatment engagement and retention. Specific Aim 2: To evaluate the impact of MOMCare on maternal clinical symptoms and functional outcomes. Specific Aim 3: To conduct an incremental cost-effectiveness analysis for a health care and welfare agency perspective that includes a) tracking the medical costs of health service use in MOMCare and usual care patients; b) monitoring the use of infant preventative health services in both groups; and c) tracking the percentage of women on Medicaid and the percentage working in both groups.

The intervention will be assessed through a practical randomized controlled trial in which we have recruited 168 pregnant women with major depression and/or dysthymia who were on Medicaid and/or received Maternal Support Services (MSS) in selected public health centers in Seattle - King County (PHSKC). Patients who were eligible and consented to study enrollment were randomly assigned to either usual care (UC) or MOMCare. Baseline and four follow-up assessments (3 - 18 months post-baseline) are scheduled for study participants in both groups. The MOMCare intervention includes a choice of brief interpersonal psychotherapy or collaborative management of antidepressant medication. Treatment response will be monitored, and the treatment will be adjusted as necessary (adding treatments, increasing dosages).

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* pregnant: 12-32 weeks gestation
* able to speak English
* telephone access
* major depressive disorder or dysthymia
* on Medicaid
* receiving health care in King County, Washington

Exclusion Criteria:

* currently in psychotherapy
* currently receiving pharmacotherapy from a psychiatrist
* high suicide risk
* history of bipolar disorder
* history of schizophrenia
* substance use or dependence in previous 3 months
* currently in a relationship with severe interpersonal violence
* history of repetitive self-harm behavior

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-01; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
SCL-20 depression | baseline, 3, 6 12, 18 month follow-ups

SECONDARY OUTCOMES:
Maternal health services utilization use and estimated costs | baseline, 3, 6 12, 18 month follow-ups
Pregnancy, delivery, birth outcomes | 6 month follow-up
Child services & outcomes (immunizations, well-child visits) | 6, 12, 18 month follow-ups
Depression free days & Quality Adjusted Life Years (EuroQol) | 3, 6, 12, 18 month follow-ups
Quality of depression care process | 3, 6, 12, 18 month follow-ups
Number of depression treatment sessions attended | 3, 6, 12, 18 month follow-ups
PHQ-9 depression | screening, baseline, 3, 6, 12, 18 month follow-ups
Edinburgh Postnatal Depression Scale | baseline, 3, 6, 12, 18 month follow-ups
Social Functioning (Work & Social Adjustment, Social & Leisure, Social Support) | baseline, 3, 6, 12, 18 month follow-ups
Inventory of Functional Status After Childbirth (IFSAC) | 6, 12, 18 month follow-ups

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Grote, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Grote NK, Katon WJ, Russo JE, Lohr MJ, Curran M, Galvin E, Carson K. COLLABORATIVE CARE FOR PERINATAL DEPRESSION IN SOCIOECONOMICALLY DISADVANTAGED WOMEN: A RANDOMIZED TRIAL. Depress Anxiety. 2015 Nov;32(11):821-34. doi: 10.1002/da.22405. Epub 2015 Sep 8. PMID 26345179
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219
- [Derived] Grote NK, Katon WJ, Russo JE, Lohr MJ, Curran M, Galvin E, Carson K. A Randomized Trial of Collaborative Care for Perinatal Depression in Socioeconomically Disadvantaged Women: The Impact of Comorbid Posttraumatic Stress Disorder. J Clin Psychiatry. 2016 Nov;77(11):1527-1537. doi: 10.4088/JCP.15m10477. PMID 28076671
- [Derived] Grote NK, Katon WJ, Lohr MJ, Carson K, Curran M, Galvin E, Russo JE, Gregory M. Culturally relevant treatment services for perinatal depression in socio-economically disadvantaged women: the design of the MOMCare study. Contemp Clin Trials. 2014 Sep;39(1):34-49. doi: 10.1016/j.cct.2014.07.001. Epub 2014 Jul 10. PMID 25016216